CLINICAL TRIAL: NCT04670224
Title: Efficiency of the Quadratus Lumborum Block for Post-operative Analgesia in Abdominoplasty Surgery
Acronym: QLB
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire, Amiens (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PI2020_843_0094
Record Dates: First submitted 2020-12-01; First posted 2020-12-17 (Actual); Last update posted 2025-05-29 (Actual); Status verified 2025-05

CONDITIONS: Quadratus Lumborum Block; Abdominoplasty; Analgesia; Locoregional Anesthesia
Keywords: Quadratus lumborum block; Abdominoplasty; Analgesia; Locoregional Anesthesia
MeSH Terms: conditions — Agnosia | interventions — Anesthesia, Intravenous

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- QLB technique (Experimental)
  Interventions: Other: QLB anesthesia
- Intravenous anesthesia without QLB (Active Comparator)
  Interventions: Other: Intravenous anesthesia without QLB

INTERVENTIONS:
Other: QLB anesthesia — The QLB is a bilateral locoregional anesthesia technique, performed after surgery, under general anesthesia and in right and then left lateral decubitus.
  Arms: QLB technique
Other: Intravenous anesthesia without QLB — only intravenous anesthesia
  Arms: Intravenous anesthesia without QLB

SUMMARY:
Abdominoplasty is a common surgical procedure in plastic surgery which causes postoperative pain and may delay patients' recovery. Surgery is potentially associated with a number of postoperative complications, whether cardiovascular, respiratory, infectious, thromboembolic, or digestive … Although they do not inevitably lead to a life-threatening prognosis, in many cases these complications delay post-operative recovery. Defined in the 1990s by Professor Henry Kehlet's Danish team, rapid rehabilitation after planned surgery is an approach to overall patient care that aims to rapidly restore previous physical and mental capacities and thus significantly reduce mortality and morbidity. Pain management is at the heart of this program and local anesthesia techniques are at the heart of early rehabilitation programs.

Described for just over a decade, Quadratus Lumborum Block (QLB) have shown their effectiveness for analgesia in abdominal, or orthopedic, or obstetrical surgery. Considering the anatomical territory concerned, this locoregional anesthesia technique seems to be very interesting in abdominoplasty to allow early rehabilitation of the patient.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients admitted for programmed dermo-lipectomy surgery with or without associated liposuction.

Exclusion Criteria:

* Pregnant woman
* Patient under 18 years of age
* Subject under guardianship or curators
* Patient allergic to local anesthetics
* Infection at the puncture sites
* Patient on morphine analgesic over the long term
* Patient on antidepressants for neuropathic pain.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 286 (Estimated)
Dates: Start 2021-03-16 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2026-01 (Estimated)

PRIMARY OUTCOMES:
Variation from baseline of morphine consumption | 24 hours after surgery

SECONDARY OUTCOMES:
Variation from baseline of morphine consumption | 1 hour after surgery
Variation from baseline of morphine consumption | 2 hours after surgery
Variation from baseline of morphine consumption | 48 hours after surgery

CONTACTS AND LOCATIONS:
Locations (1):
- BAR, Amiens, France

IPD SHARING:
Plan to Share IPD: No